CLINICAL TRIAL: NCT01940549
Title: Transcranial Direct Current Stimulation (tDCS) Enhancement of Trauma-focused Therapy for Posttraumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Director, Division of Research & Development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-13-TH-334-CTIL
Record Dates: First submitted 2013-09-02; First posted 2013-09-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: PTSD; tDCS; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trauma Focused Therapy + Sham tDCS (Sham Comparator): Trauma Focused Therapy will be conducted during the delivery of sham Transcranial Direct Current Stimulation
  Interventions: Device: Trauma Focused Therapy + tDCS
- Trauma Focused Therapy + active tDCS (Active Comparator): Trauma focused therapy will be conducted while active Transcranial Direct Current Stimulation is applied
  Interventions: Device: Trauma Focused Therapy + tDCS

INTERVENTIONS:
Device: Trauma Focused Therapy + tDCS
  Other Names: DC-STIMULATOR PLUS (neuroConn GmbH, serial 0118)

SUMMARY:
The purpose of this study is to test whether transcranial direct current stimulation (tDCS) can enhance the clinical efficacy of trauma-focused therapy for posttraumatic stress disorder.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a debilitating, often-chronic psychiatric condition emerging following a severe traumatic event. Trauma-focused therapy techniques, and primarily Prolonged Exposure, constitute the primary first-line treatment. While effective to some degree, these methods have several substantial shortcomings, including limited patient compliance (long process) and responsiveness, sustained therapeutic effect, and susceptibility to spontaneous symptom relapse. Thus, there is a considerable need for enhancing the efficacy of PTSD treatment.

Dominant theories in the field of PTSD emphasize a key role for threat-related learning and memory processes in the underlying etiology and maintenance of PTSD symptoms, such as absent or insufficient extinction of learned fear associations. Indeed, trauma-focused therapy protocols typically involve repeated imaginal or in vivo recall of traumatic memories in a systematic, controlled manner, while employing anxiety-reducing techniques, and without experiencing additional external trauma. Thus, these therapies parallel cue-extinction training within a model of learning and unlearning of conditioned responses, with the patient's diminished fear response over successive extinction trials reflecting the weakening of trauma-induced associations between the fear-provoking stimuli and the conditioned fear response. Extinction of fear responses is thus generally assumed to be one the most important underlying mechanisms of exposure therapy. Noting the limited efficacy of trauma-focused treatment (and in particular the spontaneous relapse), there is much room for improving the effectiveness of this cue-extinction process in a manner that is not dangerous to the patient (cf. extinction-enhancing pharmacological agents that are also toxic).

Transcranial direct current stimulation (tDCS) is a safe method to induce weak transcranial currents (up to 1-2 milliampere). Using 2 rubber electrodes positioned on the scalp, tDCS can be used to manipulate localized brain excitability via membrane polarisation: cathodal stimulation hyperpolarises, while anodal stimulation depolarises the resting membrane potential, whereby the induced after-effects depend on polarity, duration and intensity of the stimulation.

The investigators believe that the therapeutic efficacy of PTSD treatment can be enhanced by employing tDCS during the therapeutic process. That is, tDCS's modulatory effects on existing brain activity may enable us to render the therapeutic mechanisms operating during trauma-focused therapy more effective, leading to a more efficient and efficacious therapeutic process in terms of greater symptom reduction, greater long-term sustainability, a shorter treatment course, and broader compliance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PTSD
* Adequate physical health, including vision and hearing

Exclusion Criteria:

* Non-trauma-related major psychiatric/neurological disorder
* History of seizures, fainting spells, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or family history of treatment resistant epilepsy
* Any metal in the brain, skull or elsewhere.
* Pregnancy
* Any medical devices (i.e. Cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator)
* Intracranial lesions
* Substance abuse or dependence within the past six months
* Other criteria for MRI/tDCS

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms - Clinician Administered PTSD Scale (CAPS) | One week before treatment start (baseline measure), and up to 4 weeks after treatment end (post measure)
  Change in Clinician Administered PTSD Scale (CAPS) score from baseline to post-treatment

SECONDARY OUTCOMES:
Change in depression symptoms - Beck Depression Inventory (BDI) | One week before treatment start (baseline measure), and up to 4 weeks after treatment end (post measure)
  Change in depression severity (measure using Beck Depression Inventory (BDI)) - from baseline to post-treatment.
Change in trait anxiety symptoms - State-Trait Anxiety Inventory (Trait subscale (STAI-Trait)) | One week before treatment start (baseline measure), and up to 4 weeks after treatment end (post measure)
  Change in STAI-Trait scores - from baseline to post-treatment
Change in state anxiety symptoms - State-Trait Anxiety Inventory (State subscale (STAI-S)) | from baseline to post-treatment
  Change in STAI-State score - from baseline to post-treatment
Change in subjective quality of life - the World Health Organization Quality of Life questionnaire (WHOQOL-BREF) | One week before treatment start (baseline measure), and up to 4 weeks after treatment end (post measure)
  Change in WHOQOL-BREF scores - from baseline to post-treatment
Change in global functioning - Global Assessment of Functioning scale (GAF) | One week before treatment start (baseline measure), and up to 4 weeks after treatment end (post measure)
  Change in GAF scores - from baseline to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Talma Hendler, Prof., Principal Investigator — Tel-Aviv Sourasky Medical Center; Yair Bar-Haim, Prof., Study Director — Tel Aviv University
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel